CLINICAL TRIAL: NCT03835429
Title: Oropharynx-Brainstem-Heart Connection: A Controlled Clinical Trial to Assess Atrial Fibrillation Attenuation in Patients Treated With Oral Appliance Therapy
Brief Title: Effect of Oral Appliance Therapy on Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties.
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Emet D. Schneiderman, PhD, Professor, Biomedical Sciences, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2018-0954
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
Keywords: oral appliance; atrial fibrillation; sleep apnea; mouth shield; snoring
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Intervention Model Description: Non-randomized clinical controlled trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MyTAP oral appliance plus mouth shield (Experimental): MyTAP plus mouth shield
  Interventions: Device: MyTAP oral appliance plus mouth shield

INTERVENTIONS:
Device: MyTAP oral appliance plus mouth shield — The midline traction oral appliance (MyTAP, Airway Management Inc.(AMI), Dallas Texas) is currently marketed as a medical device to treat snoring and obstructive sleep apnea and is FDA cleared.
  Other Names: Oral appliance midline traction

SUMMARY:
This pilot study is expected to determine the efficacy of using the midline traction designed MyTAP plus mouth shield (MyTAP + MS) oral appliance combination in decreasing the number of Atrial Fibrillation events. The MS is a patient comfort accessory to the MyTAP.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is highly prevalent in the U.S. and possesses a greater risk in patients with sleep disordered breathing (SDB) versus patients without SDB. AF recurrence after catheter ablation is associated with 25% increased risk in patients with obstructive sleep apnea (OSA). One hypothesis suggests that the repeated hypoxic episodes time-linked to OSA and central sleep apnea may act as chemo-reflex triggers that enhances brainstem sympathetic activity in conjunction with responses to OSA-event hypoxia. This hypothesis is believed to induce tachycardia and cardiovascular stress. In an animal model, episodes of hypoxia were shown to induce pulmonary vein burst firing and reduction of the negative tracheal pressure promptly restored normal sinus rhythm. The Trigemino-cardiac reflex hypothesis implicates chemo- and mechanoreceptors in the oronasal cavity that provides signaling to the reticular formation via the mesencephalic nucleus of the trigeminal nerve and serves to control breathing, cardiac function, blood pH (acidity), amongst other body functions.

The sympathetic system in patients with OSA syndrome is considered to be chronically hypersensitized. A hyperarousal state suggests AF patients with OSA would tend to have AF occur more frequently in conjunction with apnea hypopnea events. An increase in autonomic sympathetic cardiac dominance with a withdrawal of cardiac parasympathetic control could easily be driven by mechanoreceptors in the oropharynx upon airway narrowing and present as decreased heart rate variability. Considering that the upper airway is often the site of greatest airflow restriction (i.e. snoring), a potential sudden rise in autonomic sympathetic nerve activity in sensory afferent fibers from the oropharynx should be the first to communicate the airflow reduction to brainstem. This theory is supported by the investigators' preliminary data and those in other reports. Oral appliance (OA) therapy that prevents snoring in conjunction with a mouth shield should simultaneously facilitate an open airway and prevent mouth breathing. The combination effect is expected to decrease vagus nerve motor efferent activity to the esophagus, facilitate nasal breathing, reduce sympathetic tone, promote stable sleep and increase HRV(heart rate variability). In patients with AF, the MyTAP + MS intervention is likely to also facilitate putatively effective medical therapies, reduce noxious AF triggers, and maintain normal oral bacterial flora levels and cardiac functioning.

ELIGIBILITY:
Inclusion Criteria:

* Pre-qualified for ablation AF intervention
* AF > 1 documented episode in a 24-hour electrocardiogram (ECG) Holter examination or implanted AF monitor in the previous 1 month prior to study enrollment; [AF episode defined as at least 12 hours duration]
* At least 8 teeth per arch to support OA device
* Use of continuous positive air pressure (CPAP)therapy and willingness to switch to OA use
* Willing and able to provide verbal and written informed consent
* Ability to understand how to apply and utilize the sleep recorder and the OA device

Exclusion Criteria:

* Patients with implantable cardiac rhythm device [pacemakers or internal cardiac device (ICDs)] or cardiopulmonary disease [heart failure, Chronic obstructive pulmonary disease (COPD), ventricular dysrhythmia]
* Unable or unwilling to complete the study demands and schedule
* Comorbidities of other sleep disorders other than OSA
* No active temporomandibular joint disorders (TMD) or jaw muscle pain, or morphological airway abnormalities
* Pre-existing difficulty swallowing; throat or neck related health issues; endocrine dysfunction; severe psychiatric and neurological disorders; intellectually disabled; handicaps limiting sleep position
* Previous OA therapy or restrictions in jaw opening
* Prior ablation of AF, myocardial infarction (MI), stroke or decompensation of heart failure within the last six months, untreated overt hyper- or hypothyroidism
* Commencement of new anti-arrhythmic drug since last monitor check
* Pharmacological dependency
* Concomitant use of hypnotic agents or other sleep aids, nicotine or alcohol intake
* Mallampati score > III
* Palatine tonsils - grade > 2
* History of Uvulopalatopharyngoplasty (UPPP) surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
AF incidence | 1 month
  Measured (%) incidence of paroxysmal AF episodes >10 seconds in duration, 1-month after starting OA (T1) therapy compared with 1-month prior to using OA.
Periodontal conditions | 1 month
  Periodontal conditions (defined according to classification developed by Centers for Disease Control and Prevention and the American Academy of Periodontology (CDC-AAP)) 24 assessment at (T0) before MyTAP + MS initiation and after 1-month (T1).

SECONDARY OUTCOMES:
MyTAP advancement change from T1 to T2 | 1 month
  OA advancement in mm
Heart rate variability analysis after 1 month compared with baseline (T0) | 1 month
  HRV in ms
Apnea hypopnea index after 1 month (T2) compared with T0-1 | 1 month
  Number of apneas and hypopneas per hour of recording
Oxygen desaturation index after 1 month (T2) compared with T0-1 | 1 month
  Percent oxygen desaturation
Epworth Sleepiness Scale (ESS); Score ≥10 is sleepy, ≥ 18 is very sleepy. | 1 month
  Change in subjective ESS score pre-OA intervention vs. after 4-weeks of OA use

CONTACTS AND LOCATIONS:
Overall Officials: Emet Schneiderman, PhD, Principal Investigator — TAMHSC
Locations (1):
- Texas A&M School of Dentistry, Health Science Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No